CLINICAL TRIAL: NCT06725784
Title: Feasibility and Cost of Robot-assisted Upper Limb Rehabilitation with Different Levels of Supervision: an Interventional Study
Brief Title: Feasibility and Cost of Robot-assisted Upper Limb Rehabilitation with Different Levels of Supervision
Acronym: RHB Clinic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Clinica Hildebrand Brissago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RHB Clinic
Record Dates: First submitted 2024-11-28; First posted 2024-12-10 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Upper Limb Sensorimotor Deficits
Keywords: unsupervised therapy; robot-assisted rehabilitation; stroke; neurorehabilitation; orthopaedic rehabilitation; upper limb rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ReHandyBot (Experimental): The therapy sessions with ReHandyBot (e.g., frequency, duration) will be scheduled based on the therapist's instruction and may vary between patients, depending on their specific needs.
  Interventions: Device: ReHandyBot

INTERVENTIONS:
Device: ReHandyBot — The ReHandyBot is a platform for hand rehabilitation with two degrees of freedom, namely forearm pronation/supination and finger flexion/extension. This device allows performing exercises targeting somatosensation and motor functions. Different exercises are implemented using virtual reality and haptic feedback; the interaction forces between subjects and ReHandyBot are measured by force sensors in the handles, allowing the control of a virtual hand and the physical interaction with the virtual environment. Mechanical properties (e.g., size, stiffness) of the objects displayed in the virtual environment are rendered by the motion/force of the instrumented handles. The type and difficulty level of the exercises are patient-specific and are automatically adapted throughout the therapy.
  The duration and frequency of the therapy sessions with ReHandyBot depend on the specific patient's needs and are set according to the therapist's instructions.

SUMMARY:
Upper limb impairments are often a result of neurological or traumatic injuries (e.g., stroke, traumatic brain injuries). These impairments may decrease independence in performing activities of daily living, severely affecting patients' quality of life. Growing evidence shows that increasing upper limb therapy dose for patients could improve functional outcomes and prevent their long-term deterioration. However, due to limited resources (e.g., the number of therapists) and high rehabilitation-related costs, providing a higher therapy dose to patients is challenging, both in the clinic and after discharge, and finding new models of care is therefore critical.

Minimally supervised or unsupervised robot-assisted therapy (i.e., patients training with rehabilitation devices with minimal to no supervision of an external person) holds the promise of allowing an increase in therapy dose with little impact on the additional resources needed. Because of their ability to provide active support and measure a wide set of parameters, actuated (active) rehabilitation robots seem to be the best solution for this therapy setting. However, such devices are often complex to use and have never been extensively tested minimally or unsupervised. Consequently, the data available on their feasibility and cost-effectiveness is limited.

At the Rehabilitation Engineering Laboratory (RELab, ETH Zurich), we developed ReHandyBot, an actuated device for unsupervised upper limb therapy. The device has already been tested with stroke patients in an unsupervised setting, with positive results regarding usability and increase in therapy dose. The main goal of this project is, therefore, to investigate the feasibility and cost of our robot-assisted continuum of care model (i.e., from inpatient to ambulatory). Specifically, we aim to evaluate the feasibility of integrating ReHandyBot into the clinical routine and perform a preliminary cost-benefit analysis of supervised, minimally supervised, and unsupervised robot-assisted therapy. Furthermore, we will also gather data on the overall dose of robot-assisted therapy and the intensity of use of the device in a clinical and ambulatory setting.

DETAILED DESCRIPTION:
The ReHandyBot is a platform for hand rehabilitation with two degrees of freedom, namely forearm pronation/supination and finger flexion/extension. This device allows performing exercises targeting somatosensation and motor functions. Different exercises are implemented using virtual reality and haptic feedback; the interaction forces between subjects and ReHandyBot are measured by force sensors in the handles, allowing the control of a virtual hand and the physical interaction with the virtual environment. Mechanical properties (e.g., size, stiffness) of the objects displayed in the virtual environment are rendered by the motion/force of the instrumented handles. The type and difficulty level of the exercises are patient-specific and are automatically adapted throughout the therapy.

The duration and frequency of the therapy sessions with ReHandyBot depend on the specific patient's needs and are set according to the therapist's instructions.

The main goals of this study are to:

(i) Evaluate the feasibility of integrating ReHandyBot into the routine of rehabilitation clinics and ambulatories.

(ii) Perform a cost-benefit analysis of supervised, minimally supervised, and unsupervised therapy with the device.

The secondary goals are to investigate:

(iii) The intensity of use of ReHandyBot by the facilities. (iv) The increase in therapy dose for the patients using the device minimally or unsupervised compared to usual care.

(v) The quantity and characteristics of patients who can train supervised, minimally, or unsupervised with the device.

(vi) Usability and user experience.

All the patients admitted to the clinic or ambulatory will be screened for participation in this study. Eligible patients will receive robot-assisted therapy sessions with the ReHandyBot in parallel to their conventional therapy program. During therapy with ReHandyBot, the patient sits comfortably on a chair in front of a screen and places the fingers of the impaired hand on the handles of the device.

The eligibility of the patients will be checked during the admission visit, after which, for eligible patients, a trial session with ReHandyBot will be scheduled. During the trial session, the supervising therapist will decide if the patient can really benefit from training with ReHandyBot, and if yes, the therapist will integrate supervised therapy sessions with the device into the therapy schedule of the patient. Then, during the supervised sessions, the therapist will use a checklist to decide if a patient can train minimally supervised (i.e., group sessions) or unsupervised. If this will be the case, the minimally or unsupervised therapy sessions will be added to the therapy schedule of the patient. The therapy sessions with ReHandyBot (e.g., frequency, duration) will be scheduled based on the therapist's instruction and may vary between patients, depending on their specific needs. On the day of the last session with ReHandyBot, patients will fill in questionnaires to rate its usability and user experience.

For each recruited patient, data regarding demographics, medical condition, clinical and cognitive assessments, therapy dose, and device data will be recorded on the CRF. Medical and assessment data will be data routinely collected at the clinic and ambulatory. We will not perform evaluations specifically for this study.

At the end of the study, data regarding costs, intensity of use, and device retention will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject.
* Female and male patients between 18 and 90 years old
* Presence of an upper limb deficit derived from any disease or event that, according to the responsible clinicians, could be improved by therapy with ReHandyBot.

Exclusion Criteria:

* Pathologies that may interfere with the training with ReHandyBot.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-04 (Estimated); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Cost of ReHandyBot | Monitored through study completion (expected duration: 5 years).
  Manufacturing costs of ReHandyBot and cost of its maintenance over the duration of the study in Swiss Francs (CHF). These costs are monitored by the manufacturer.
Cost of the clinical staff supporting therapy with ReHandyBot | Monitored through study completion (expected duration: 5 years).
  Cost in Swiss Francs related to the clinical staff being present during the therapy sessions with ReHandyBot. This will be extrapolated from the software that the clinic uses to handle the schedules of the therapists. This cost is calculated by multiplying the number of therapy sessions with the device performed by the therapists of the clinic by the hourly rate of the therapists.
Number of supervised therapy sessions with ReHandyBot | Monitored through study completion (expected duration: 5 years).
  Number of therapy sessions with ReHandyBot performed by the participants under the supervision of a therapist (i.e., 1-to-1 therapy sessions). This number is extrapolated from the software that the clinic uses to handle the schedules of the patients.
Number of minimally supervised therapy sessions with ReHandyBot | Monitored through study completion (expected duration: 5 years).
  Number of therapy sessions with ReHandyBot performed by the participants under minimal supervision of a therapist (e.g., group sessions). This number is extrapolated from the software that the clinic uses to handle the schedules of the patients.
Number of unsupervised therapy sessions with ReHandyBot | Monitored through study completion (expected duration: 5 years).
  Number of therapy sessions with ReHandyBot performed by the participants without the supervision of a therapist (i.e., the therapist is not present). This number is extrapolated from the software that the clinic uses to handle the schedules of the patients.
Patient-to-therapist ratio of the therapy sessions with ReHandyBot | Monitored through study completion (expected duration: 5 years).
  Ratio of the number of patients to number of therapists present during the therapy sessions with ReHandyBot, where a higher ratio (i.e., multiple patients for one therapist) constitutes an economic benefit for the clinic. This ratio is extrapolated from the software of the clinic handling the schedules of patients and therapists.

SECONDARY OUTCOMES:
Feasibility of integrating ReHandyBot into the routine of a rehabilitation clinic: adverse events | Monitored through study completion (expected duration: 5 years).
  Feasibility of integrating ReHandyBot into the routine of a rehabilitation clinic assessed as the number of adverse events related to the device.
Feasibility of integrating ReHandyBot into the routine of a rehabilitation clinic: device deficiencies | Monitored through study completion (expected duration: 5 years).
  Feasibility of integrating ReHandyBot into the routine of a rehabilitation clinic assessed as the number of device deficiencies.
Feasibility of integrating ReHandyBot into the routine of a rehabilitation clinic: usage | Monitored through study completion (expected duration: 5 years).
  Feasibility of integrating ReHandyBot into the routine of a rehabilitation clinic assessed as the usage (i.e., number of therapy sessions) of the device over time (i.e., if the device is no longer used after a short period, it means that it was not feasible to integrate it into the clinical routine of patients and therapists).
Intensity of use of ReHandyBot | Monitored through study completion (expected duration: 5 years).
  Intensity of use of ReHandyBot, assessed as the number of hours per day when the device is occupied by a patient.
Increase in therapy dose: minutes | From participant's recruitment (day 0) until discharge from the clinic (on average: after 4 weeks).
  The increase in therapy dose in minutes for the patients using ReHandyBot minimally or unsupervised compared to usual care.
Increase in therapy dose: percentage | From participant's recruitment (day 0) until discharge from the clinic (on average: after 4 weeks).
  The increase in physical therapy dose in percentage for the patients using ReHandyBot minimally or unsupervised compared to usual care.
Quantity of patients training with ReHandyBot | Monitored through study completion (expected duration: 5 years).
  Quantity of patients training with ReHandyBot expressed as the percentage of patients training with the device out of the total patients admitted to the clinic.
Characteristics of patients training with ReHandyBot | Monitored through study completion (expected duration: 5 years).
  Characteristics (e.g., age, diagnosis) of patients training with ReHandyBot compared to the patients who are not eligible or able to train with ReHandyBot.
Reason why patients eventually stop training with ReHandyBot | From participant's recruitment (day 0) until the last session performed with the device (on average: 4 weeks).
  Reason why an eligible patient eventually stops training with the device (e.g., due to not liking the device).
Evolution of patient's satisfaction with robot-assisted therapy as assessed by a 5-point scale | Monitored over the whole protocol duration (i.e., from the first to the last therapy session with ReHandyBot, on average 4 weeks).
  A 5-point scale is presented by the robot at the end of each therapy session to measure patient's satisfaction with robot-assisted therapy.
Usability as assessed by the System Usability Scale | Measured after two weeks from the first therapy session with ReHandyBot performed by a participant.
  Usability of the ReHandyBot measured with the System Usability Scale. The possible response options vary between 1 (strongly disagree) and 5 (strongly agree).
User experience - Net Promoter Score | Measured after two weeks from the first therapy session with ReHandyBot performed by a participant.
  The Net Promoter Score consists of the question "How likely would you be to recommend therapy with ReHandyBot to another patient?". The possible response options vary between 1 (extremely unlikely) and 10 (extremely likely).

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Clinica Hildebrand Centro di riabilitazione Brissago, Brissago
  - Clinica Hildebrand Centro Ambulatoriale Lugano, Lugano

IPD SHARING:
Plan to Share IPD: No